CLINICAL TRIAL: NCT01191580
Title: Interpersonal Therapy for Depression in Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #5996/7033R
Record Dates: First submitted 2010-06-24; First posted 2010-08-31 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Interpersonal Psychotherapy (Experimental): Interpersonal Psychotherapy is a brief, manualized therapy that has shown efficacy in treating major depression in several controlled trials including a large trial for depressed HIV-infected individuals and other randomized trials in depressed individuals with other comorbid medical illnesses. Research shows that Interpersonal Psychotherapy improves social skills and functioning. Interpersonal Psychotherapy has shown remarkable flexibility and efficacy across age ranges, cultures, formats, and modes of delivery. We recently obtained promising pilot data in a small open trial on the acceptability and efficacy of individual IPT for depressed breast cancer patients of diverse ethnic background, socioeconomic status, and cancer progression stage.
  Interventions: Behavioral: Interpersonal Psychotherapy
- Problem-Solving Therapy (Experimental): Problem-Solving Therapy is a brief, manualized form of cognitive-behavioral therapy (CBT) that has been adapted to treat depression in cancer patients, and has shown highly promising results.
  Interventions: Behavioral: Problem-Solving Therapy
- Brief Supportive Psychotherapy (Active Comparator): Brief Supportive Psychotherapy, a relatively unstructured psychotherapy commonly used in clinical practice, focuses on the patient's affect. It builds a strong therapeutic alliance through careful, empathic listening and validating and encouraging toleration of the patient's emotions. It has shown promising results in depressed individuals with cancer and other medical illnesses.
  Interventions: Behavioral: Brief Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — Interpersonal Psychotherapy will consist of twelve 50-minute sessions delivered within a period of 16 weeks. IPT is divided into three phases.
  Other Names: IPT
  Arms: Interpersonal Psychotherapy
Behavioral: Problem-Solving Therapy — Problem-Solving Therapy will also consist of 12 50-minute sessions. The goals of the PST are: 1) to assist patients to identify and link life situations related to the depression; 2) to increase the effectiveness of the patient's problem-solving attempts at coping with current problems based on an intervention carried out in a concrete, structured and, unambiguous manner.
  Other Names: PST
  Arms: Problem-Solving Therapy
Behavioral: Brief Supportive Psychotherapy — The treatment approach will follow the standard supportive therapy approaches used in depression and medical illness, as noted below.
  Brief Supportive Psychotherapy has a biopsychosocial perspective, recognizing contributions of genetic predisposition and neuroendocrine factors (Novalis et al., 1993, p. 257-277). Its goals are to maximize patient function during crisis, to support the patient's judgment with the therapist's reasoning skills, and to engender hope for recovery. Primary techniques and practices include reality testing; being relatively accepting of existing defenses but attempting to restructure them when appropriate; and, using self-esteem enhancing measures.
  Other Names: BSP
  Arms: Brief Supportive Psychotherapy

SUMMARY:
The investigators propose a randomized clinical trial to compare the efficacy of Interpersonal Psychotherapy (IPT), Problem-Solving Therapy (PST), and Brief Supportive Psychotherapy (BSP), in improving depressive symptoms, psychosocial functioning, and quality of life among patients with breast cancer and major depressive disorder (MDD).

DETAILED DESCRIPTION:
Depressive symptoms and disorders are common in cancer patients: up to 58% have depressive symptoms, and 38% meet Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria for major depressive disorder (MDD). Depression worsens over the course of cancer treatment, persists long after cancer therapy, recurs with recurrence of cancer, and negatively affects patients' adherence to cancer treatment, survival, symptom management, psychosocial functioning, and quality of life. As surviving cancer becomes increasingly common, there is an urgent need to establish an empirical basis for the provision of evidence-based treatments to depressed cancer patients.We propose a randomized clinical trial to compare the efficacy of Interpersonal Psychotherapy (IPT), Problem-Solving Therapy (PST), and Brief Supportive Psychotherapy (BSP), in improving depressive symptoms, psychosocial functioning, and quality of life among patients with breast cancer and major depressive disorder. The study is based on several complementary observations from recent studies. First, 30-60% of cancer patients experience clinically significant depressive symptoms. Second, depression is associated with poorer cancer outcomes. Third, over the course of the illness, depression recurs or persists for a significant number of cancer patients. Fourth, several recent reviews have indicated that, despite decades of research and hundreds of studies, the available evidence is insufficient to empirically guide the treatment of major depressive disorder in cancer patients. This has led the national institute of health, the Institute of Medicine, and other experts to call for well-designed, controlled trials of the treatment of depression in cancer patients.

Interpersonal Psychotherapy is a brief, manualized therapy that has shown efficacy in treating major depression in several controlled trials including a large trial for depressed HIV-infected individuals and other randomized trials in depressed individuals with other comorbid medical illnesses. Research shows that Interpersonal Psychotherapy improves social skills and functioning. Interpersonal Psychotherapy has shown remarkable flexibility and efficacy across age ranges, cultures, formats, and modes of delivery. We recently obtained promising pilot data in a small open trial on the acceptability and efficacy of individual Interpersonal Psychotherapy for depressed breast cancer patients of diverse ethnic background, socioeconomic status, and cancer progression stage. Problem-Solving Therapy is a brief, manualized form of cognitive-behavioral therapy (CBT) that has been adapted to treat depression in cancer patients, and has shown highly promising results. Brief Supportive Psychotherapy, a relatively unstructured psychotherapy commonly used in clinical practice, focuses on the patient's affect. It builds a strong therapeutic alliance through careful, empathic listening and validating and encouraging toleration of the patient's emotions. It has shown promising results in depressed individuals with cancer and other medical illnesses.

ELIGIBILITY:
Inclusion Criteria:

* A primary psychiatric diagnosis of Major Depressive Disorder as defined by: a score of 18 or above in the 17-item Hamilton Depression Scale; Male or female ages 18+;
* Ability to give consent
* Diagnosis of Breast Cancer
* Patients may be either English or Spanish speaking

Exclusion Criteria:

* Lifetime history of psychosis or bipolar disorder
* Patients meeting diagnostic statistic manual for mental disorder criteria for alcohol or substance use disorders who require acute detoxification.
* Current suicide risk.
* Advanced cancer or other condition that limits remaining life expectancy to less than 6 months.
* Patients who are receiving effective medication for Depression

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-10; Primary Completion 2016-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAMD-17) | week 12
  Change in HAMD-17 following acute treatment is the primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: John C. Markowitz, M.D., Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided